CLINICAL TRIAL: NCT01182857
Title: Quality of Life and Neuropsychiatric Sequelae in Patients Treated With Gene Therapy for ADA-SCID and in Their Parents
Status: Withdrawn | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100151; 10-HG-0151
Record Dates: First submitted 2010-08-14; First posted 2010-08-17 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2014-09-25

CONDITIONS: ADA-SCID
Keywords: Quality of Life; Gene Therapy; ADA-SCID; SCID-ADA; Severe Combined Immunodeficiency
MeSH Terms: conditions — Severe combined immunodeficiency due to adenosine deaminase deficiency; Severe Combined Immunodeficiency

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

* Severe combined immunodeficiency (SCID) is a rare inherited disorder in which certain white blood cells have impaired function and are unable to properly fight infections. SCID typically appears within the first year of life and is characterized by multiple, recurrent severe infections. More than 10 percent of all cases of SCID involve a deficiency of an enzyme called adenosine deaminase (ADA), and these SCID patients also tend to have impaired brain function or psychiatric disorders. Researchers are attempting to treat ADA-SCID patients with an experimental gene therapy, and a research protocol has been established for those who are participating in this therapy.
* Little is known about quality of life in individuals with ADA-SCID, but researchers believe that the effects of the disease and the treatments may cause a decreased quality of life in both patients and their parents. Another potential cause of decreased quality of life in ADA-SCID is the associated psychiatric and neurological problems caused by the disease. Researchers are interested in studying quality of life in individuals with ADA-SCID and their parents to provide more information about the disease.

Objectives:

* To evaluate whether gene therapy alters the quality of life or neuropsychiatric status of children with ADA-SCID.
* To monitor for intellectual, attention, memory, or specific learning disorders in children with ADA-SCID.
* To evaluate whether undergoing gene therapy has an effect on parenting stress of parents whose children have ADA-SCID.

Eligibility:

* Children who are participating in the ADA-SCID gene therapy research protocol (01-HG-0189).
* Parents of children who are participating in the ADA-SCID gene therapy research protocol (01-HG-0189).

Design:

* All of the testing and questionnaires will be done in the pediatric or adult clinic.
* Participating children will have tests of intelligence, manual dexterity, reaction time, basic reading and arithmetic skills, speech, and memory. These tests will be given before the start of the therapy, and then once a year for 5 years.
* Participating children will also complete questionnaires on quality of life. These questionnaires will be given before the start of the therapy, 3 months and 6 months after the therapy, and then every 6 months for a total of 5 years.
* Additional psychological tests may be given at the discretion of the study researchers.
* Parents will complete questionnaires to provide background medical information and report on quality of life and parental stress. The background information questionnaires will be given at the start of the therapy and then once a year for 5 years, the parental stress questionnaires will be given at the start of the therapy and then every 6 months for 5 years, and the quality of life questionnaires will be given at the same time as the child quality of life questionnaires.
* This protocol is separate from the gene therapy treatment protocol.

DETAILED DESCRIPTION:
The objectives of this study are to measure quality of life, neuropsychological sequelae and parental stress before and after gene therapy for ADA-SCID. The population to be studied will include up to five patients being treated with gene therapy at the NIH Clinical Center and five of their parents. The design of the study will be a non-randomized, longitudinal psychometric evaluation. Neuropsychological outcome measures will be the following battery: Wechsler Preschool and Primary Scale of Intelligence - Third Edition (WPPSI-III) or the Wechsler Intelligence Scale for Children - Fourth Edition (WISC-IV); the Wide Range Achievement Test - Fourth Edition (WRAT-4); subtests of the NEPSY; The Expressive One Word Picture Vocabulary Test (EOWPVT); Grooved Pegboard; Continuous Performance Test (CPT); Selective Reminding Test; and the Adaptive Behavior Assessment System- Second Edition. Quality of life will be measured with the PedsQL and parental stress will be measured with the Parenting Stress Index.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients:

* Patients must be enrolled on protocol 01-HG-0189 in order to be eligible for enrollment on this protocol.
* Written informed consent from adult patients, or from the parents or guardians of minor patients must be obtained. Assent must be obtained from minor children when applicable.
* Patients must be English-speaking. Not all of the study instruments have been validated in other languages, and personnel are not available with training to administer the instruments in other languages.

Parents or Guardians

* Parents must have a child enrolled on protocol 01-HG-0189 in order to be eligible for enrollment on this protocol. Guardians must have a ward enrolled on protocol 01-HG-0189 in order to be eligible for enrollment on this protocol.
* Written informed consent must be obtained from parents or guardians.

EXCLUSION CRITERIA:

* Inability to complete the study instruments. This includes inability to speak English. Not all of the study instruments have been validated in other languages, and personnel are not available to administer the test instruments in other languages.
* Judgment of the clinical investigators that participation would be detrimental to the patient, parent or guardian.
* Judgment of the clinical investigators that participation would be detrimental to the study.

Ages: 5 Months to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2010-08-05; Study Completion 2014-09-25

PRIMARY OUTCOMES:
Quality of life and neuropsychiatric status of patients being treated with gene therapy for ADA-SCID. | 2 years

SECONDARY OUTCOMES:
Parental stress in parents of children being treated with gene therapy for ADA-SCID. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Sokolic, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)

REFERENCES:
- [Background] Varni JW, Seid M, Kurtin PS. PedsQL 4.0: reliability and validity of the Pediatric Quality of Life Inventory version 4.0 generic core scales in healthy and patient populations. Med Care. 2001 Aug;39(8):800-12. doi: 10.1097/00005650-200108000-00006. PMID 11468499
- [Background] Fasth A, Nystrom J. Quality of life and health-care resource utilization among children with primary immunodeficiency receiving home treatment with subcutaneous human immunoglobulin. J Clin Immunol. 2008 Jul;28(4):370-8. doi: 10.1007/s10875-008-9180-9. Epub 2008 Feb 7. PMID 18256911
- [Background] Abidin RR, Wilfong E. Parenting stress and its relationship to child health care. Child Health Care. 1989 Spring;18(2):114-6. doi: 10.1207/s15326888chc1802_9. PMID 10292918